CLINICAL TRIAL: NCT00946595
Title: A Study Comparing Efficacy and Tolerance of Two Maintenance Strategies : a Monotherapy With Lopinavir/Ritonavir or a Single-tablet Triple Therapy by Efavirenz/Emtricitabin/Tenofovir in HIV-1 Infected Patients With HIV RNA Below 50 cp/mL
Brief Title: Evaluation of a Lopinavir/Ritonavir Monotherapy vs a Triple Therapy as Maintenance Regimens in HIV-1 Infected Patients
Acronym: ANRS 140 DREAM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Abbott (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-009776-13; ANRS 140 DREAM
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: HIV Infections
Keywords: Undetectable; HIV infections; Monotherapy; Lopinavir/ritonavir; Protease inhibitor; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- efavirenz/emtricitabin/tenofovir (Active Comparator)
  Interventions: Drug: efavirenz/emtricitabin/tenofovir
- lopinavir/ritonavir (Experimental)
  Interventions: Drug: lopinavir/ritonavir

INTERVENTIONS:
Drug: efavirenz/emtricitabin/tenofovir — 1x600/200/245 mg per day (one tablet) between W0 et W98
  Other Names: Atripla
  Arms: efavirenz/emtricitabin/tenofovir
Drug: lopinavir/ritonavir — 4 x 200/50 mg (4 tablets) once a day between W0 and W98
  Other Names: Kaletra
  Arms: lopinavir/ritonavir

SUMMARY:
A 2-year multicenter, phase II/III, randomized active-controlled trial to evaluate the efficacy and tolerance of two maintenance strategies in HIV-1 infected patients with HIV RNA below 50 copies/mL : a monotherapy with lopinavir/ritonavir or a single-tablet triple therapy (EFV/FTC/TDF).

DETAILED DESCRIPTION:
Today, one of the challenges of HIV treatment is to overcome side effects and toxicity of long term antiretroviral therapy. A promising approach may be the simplification of treatment maintenance strategies, sparing certain antiretroviral drug classes. This is a two-year prospective phase II/III, multicenter randomized trial to evaluate the efficacy and tolerance of a lopinavir/ritonavir monotherapy as a maintenance regimen in HIV-infected adults. Enrolled patients must have had stable antiretroviral treatment and HIV-1 RNA below 50 cp/mL over the previous 12 months, and no prior treatment failure. Provided informed consent, 420 patients are randomized in a 1:1 ratio to two open-label treatment groups and receive either lopinavir/r 800/200mg per day or EFV/FTC/TDF 600/200/245 mg per day (fixed dose combination). The main objective is to assess treatment efficacy and tolerance after 2 years. In 80 patients, repeated DEXA measurements are performed during the trial in order to evaluate changes in bone mineral density and in body composition.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection
* Stable antiretroviral treatment over 6 months
* HIV-1 RNA < 50 cp/mL for at least 12 months
* Lymphocytes CD4+ > 200/mm3
* Lymphocytes CD4+ nadir > 100/mm3
* Absence of prior treatment failure (defined by two successive HIV-1 RNA ≥ 50 cp/mL under NNRTI or PI treatment)
* Absence of documentation of a mutation conferring NRTI or NNRTI resistance or a primary mutation in the protease gene
* Written informed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Woman of child bearing potential without efficient contraception
* Pregnant or breastfeeding woman
* HBV infection (HbS Ag+)
* HBC infection requiring specific treatment during the trial
* Liver cirrhosis Child-Pugh C
* HIV-1/HIV-2 Co-infection or isolated HIV-2 infection
* Ongoing interleukin or interferon treatment
* Co-administration of contraindicated treatments
* Hypersensibility to efavirenz or lopinavir/r
* Absolute neutrophil count < 750/mm3, hemoglobin < 8g/dL, platelets < 60.000/mm3, creatinine clearance < 50 mL/min, ASAT, ALAT, lipase, alkaline phosphatase or total bilirubin > 3 ULN, CD4 nadir < 100/mm3.
* Participation in another clinical trial interfering with the study drug assignment in DREAM
* Subject under legal guardianship or incapacitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without treatment failure at Week 96 | Week 96

SECONDARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA below 50 cp/mL at all time points during the trial | From Week 0 to Week 96
Proportion of patients with plasma HIV-1 RNA below 50 cp/mL at Week 96 | Week 96
Proportion of patients with plasma HIV-1 RNA below 400 cp/mL at all time points during the trial | From Week 0 to Week 96
Evolution of CD4 cell count between Week 0 and Week 96 | Between Week 0 and Week 96
Evaluation of treatment adherence | From Week 0 to Week 96
Evaluation of treatment tolerance | From Week 0 to Week 96
Number and type of new resistance mutations in case of two successive plasma HIV-1 RNA ≥ 400 cp/mL | From Week 0 to Week 96
Proportion of patients with loss of future drug options | From Week 0 to Week 96
Evaluation of quality of life assessments | From Week 0 to Week 96
Prevalence of acquired impairment in cognitive functioning, involving at least two ability domains, without interference in daily functioning or functioning complaint between Week 0 and Week 96 | Between Week 0 and Week 96
Prevalence of acquired impairment in cognitive functioning, involving at least two ability domains, with interference in daily functioning or functioning complaint between Week 0 and Week 96 | Between Week 0 and Week 96
Evolution of densitometric parameters between Week 0 and Week 96 in 80 patients | Between Week 0 and Week 96
Analysis of the determinants of the durability of the virological response | From Week 0 to Week 96
Assessment of pharmacokinetic and pharmacodynamic parameters in both groups if relevant | From Week 0 to Week 96

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales Hopital Saint-Antoine, Paris, France

REFERENCES:
- [Derived] Garay OU, Nishimwe ML, Bousmah MA, Janah A, Girard PM, Chene G, Moinot L, Sagaon-Teyssier L, Meynard JL, Spire B, Boyer S. Cost-Effectiveness Analysis of Lopinavir/Ritonavir Monotherapy Versus Standard Combination Antiretroviral Therapy in HIV-1 Infected Patients with Viral Suppression in France (ANRS 140 DREAM). Pharmacoecon Open. 2019 Dec;3(4):505-515. doi: 10.1007/s41669-019-0130-7. PMID 30968368
- [Derived] Lambert-Niclot S, Grude M, Meynard JL, Marcelin AG, Valantin MA, Flandre P, Izopet J, Moinot L, Bouteloup V, Calvez V, Katlama C, Girard PM, Morand-Joubert L. Ultrasensitive Human Immunodeficiency Virus Type 1 Viral Load as a Marker of Treatment Choice for Simplification Strategies. Clin Infect Dis. 2018 Nov 28;67(12):1883-1889. doi: 10.1093/cid/ciy382. PMID 29767684
- See also: Related Info — http://www.anrs.fr